CLINICAL TRIAL: NCT04247334
Title: Brain Circuitry of Inhibitory Control: Effects of Modulation
Brief Title: Inhibitory Control: Effects of Modulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1352651-9
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Young Adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cautious Participants (No Intervention): Participants who have low scores on a self-report of inhibitory control abilities (BRIEF-Inhibit).
- Impulsive Participants- Active Stimulation (Experimental): Participants who have high scores on a self-report of inhibitory control abilities (BRIEF-Inhibit) who are randomized to active stimulation.
  Interventions: Device: Transcranial direct current stimulation
- Impulsive Participants- Sham Stimulation (Sham Comparator): Participants who have high scores on a self-report of inhibitory control abilities (BRIEF-Inhibit) who are randomized to sham stimulation.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — 20 minutes of 2 milliamp transcranial direct current stimulation
  Arms: Impulsive Participants- Active Stimulation; Impulsive Participants- Sham Stimulation

SUMMARY:
Inhibitory control is relevant to many clinical disorders, including substance abuse/dependence, obsessive-compulsive disorder, and attention-deficit hyperactivity disorder. This proposal is designed to assess brain networks related to response inhibition in healthy young adults, and use neuromodulation to change these networks and behavioral performance on a response inhibition task. Having an understanding of the brain mechanisms involved in response inhibition may enable us to improve pre-existing treatments for disorders with inhibitory control difficulties.

ELIGIBILITY:
Inclusion Criteria:

1. Low (<1sd below the mean on the BRIEF-Inhibit) or high (>1sd above the mean on BRIEF-Inhibit scale)
2. English fluency to ensure comprehension of study measures and instructions.

Exclusion Criteria:

1. Presence of medical conditions contraindicated for tDCS, including history of any known intracranial pathology, epilepsy or seizures, traumatic brain injury, brain tumor, stroke, implanted medical devices, current pregnancy or women of childbearing age not using effective contraception, or any other serious medical conditions or health problems that would interfere with participation (e.g., skin condition)
2. Inability to undergo MRI
3. Current substance abuse disorder
4. Currently prescribed psychiatric medications.
5. Active mania or psychosis

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
fMRI connectivity at rest | 2 weeks
  Changes in resting state connectivity of the inhibitory control information
fMRI connectivity during a stop signal task | 2 weeks
  Changes in task-based connectivity on the stop signal task

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No